CLINICAL TRIAL: NCT05741255
Title: Effect of Acceptance and Commitment Therapy Based Interventions on Mental Health and Cognitive Impairment for Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1322023
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Acceptance and Commitment Therapy, Mental Health, Cognitive Impairment,Colorectal Cancer
MeSH Terms: conditions — Psychological Well-Being; Cognitive Dysfunction; Colorectal Neoplasms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): After random sampling and dividing patients into two groups of study and control. Patients from the study and control groups will be interviewed individually by the researcher to apply the study tools. Acceptance and Commitment Therapy will be carried out for patients in the study group
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Control group (Active Comparator): Those in the control group will be left without any intervention to undergo the usual unit routine care.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — type of mindful psychotherapy that helps you stay focused on the present moment and accept thoughts and feelings without judgment. It aims to help you move forward through difficult emotions so you can put your energy into healing instead of dwelling on the negative.

SUMMARY:
The present study aims to:

Determine the effect of acceptance and commitment therapy-based interventions on mental health and cognitive impairment for patients with advanced colorectal cancer.

Research Hypothesis:

Cancer patients who receive acceptance and commitment therapy-based interventions will exhibit better mental health and lower cognitive impairments than those who didn't receive it.

DETAILED DESCRIPTION:
6) Patients' medical charts in the unit will be reviewed to identify those who meet the inclusion criteria. Patients who meet the predetermined inclusion criteria will be randomly recruited in the study. After random sampling and dividing patients into two groups of study and control. Patients from the study and control groups will be interviewed individually by the researcher to apply the study tools. Acceptance and Commitment Therapy will be carried out for patients in the study group while those in the control group will be left without any intervention to undergo the usual unit routine care.

7) The researcher was undergoing a period of training on Acceptance and Commitment Therapy (ACT) through online academic training at Association for Contextual Behavioral Science (ACBS) for 8 weeks with 16 credits hours'certificate by (Harris, 2015). Before embarking on the actual study, the researcher passed through independent teaching about acceptance and commitment therapy under the direction, guidance, and supervision of the thesis supervisors. This included a discussion of the theoretical foundation of ACT as well as the accuracy and appropriateness of the exercises used and needed for each session.

8) The therapy consisted of six sessions, each session of acceptance and commitment therapy was developed based on general and specific objectives. An expert professor in the nursing education field revised the ACT sessions' overall objectives and the specific ones. The overall objectives of each session and the content of the sessions were translated into Arabic.

ELIGIBILITY:
Inclusion Criteria:

Are not participating in any type of psychotherapy, score high in the cognitive impairment questionnaire.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Mental Health Continuum-Short Form | 2 weeks
  The original 14-item Mental Health Continuum-Short was developed by (Keyes & psychology, 2004) in response to demands for a brief self-rating assessment tool that combined the three components of wellbeing: emotional, social, and psychological.
Montreal Cognitive Assessment | 2 weeks
  The one-page Montreal Cognitive Assessment (MoCA) was used to assess the eight cognitive domains of attention (6 points), visuospatial/executive functions (5 points), short-term memory (5 points), naming (3 points), language (3 points), orientation (6 points), and abstraction (2 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No